CLINICAL TRIAL: NCT00811356
Title: A Single-Blind, Placebo-Controlled, Randomized First Time in Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Dose Escalation of GSK932121 in Healthy Adult Subjects
Brief Title: A First Time in Human Study in Healthy Volunteers to Investigate a New Medicine to Treat Malaria
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: safety issues (toxicity)
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 111319
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Malaria
Keywords: Food Effect; Drug-Drug Interaction; Antimalarial; First Time In Human; Single Dose; Repeat Dose
MeSH Terms: conditions — Malaria | interventions — Rosiglitazone; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Dose, Repeat Dose, Drug-Drug Interaction (Experimental): GSK932121 or placebo will be administered as a single dose with or without food in a dose escalation manner. Once the results from the single dose is obtained and reviewed, GSK932121 or placebo will be administered as a repeat dose. The results from each repeat dose level will be reviewed prior to determining the next repeat dose level.
  To better understand the effect of GSK932121 on rosiglitazone and rosuvastatin, a drug-drug interaction arm will also be investigated in this study. Rosiglitazone and rosuvastatin will be administered alone, then GSK932121 will be given as a repeat dose. Rosiglitazone and rosuvastatin will then be administered in combination with GSK932121.
  Interventions: Drug: GSK932121; Rosiglitazone; Rosuvastatin

INTERVENTIONS:
Drug: GSK932121; Rosiglitazone; Rosuvastatin — GSK932121 is the study drug that will be tested in all parts of this study as described above. Rosiglitazone and rosuvastatin will only be tested in the drug-drug interaction substudy.

SUMMARY:
The purpose of this study is to determine if the study drug (antimalarial medication) is safe when given to healthy subjects as a single dose or as repeated doses, to understand the effect of food on single doses of study drug and to determine if the study drug has an effect on other approved medications such as rosiglitazone and rosuvastatin.

DETAILED DESCRIPTION:
Malaria is a type of parasitic infection, common in tropical and subtropical regions of the world, including parts of the Americas, Asia, and Africa. In recent years there has been a rapid spread of drug resistant malaria which makes it necessary to develop new antimalarial treatments. In animal studies, GSK932121 is shown to be able to kill the malaria parasite and is fully active against drug resistant malaria parasites. It is hoped that information collected on this study will lead to an improved treatment for malaria.

This is a first time in human fusion study which has 3 parts:

Part A - single dose escalation/ food effect: a study where the study drug is given once only- first at the lowest dose of in a group of participants and the dose increased only if the previous dose is found to be safe. It also looks at the effect of food on the study drug in the body Part B - repeat dose escalation: a study where the study drug will be given daily for up to 7 days - first at a lower dose in a group of participants and the dose increased for the next group only if the previous dose is found to be safe and Part B - drug-drug interaction: a study where the study drug will be given daily for up to 7 days at a dose determined to be safe in previous groups of participants and looking at the effect of the study drug on other specific approved medications (such as rosiglitazone--a diabetic medication and rosuvastatin--a cholesterol lowering medication) in the body.

Safety will be assessed by measurement of vital signs, cardiac monitoring, spirometry, collection of adverse event assessments, renal biomarkers and laboratory safety tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age, inclusive
* Females of non-childbearing potential (as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* Body weight > 50 kg and BMI within the range 19 - 31 kg/m2 (inclusive)
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block

Exclusion Criteria:

* Positive pre-study drug/alcohol screen
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of the study
* Participation in a clinical trial with an investigational product within 30 days or 5 half-lives of the investigational product (whichever is longer) prior to start of the new study
* Exposure to more than four new drugs or within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that would be contraindicated
* Donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or history of heparin-induced thrombocytopenia if heparin is used to maintain the patency of an intravenous cannula.
* Asthma or a history of asthma
* Smoking or history or regular use of tobacco- or nicotine-containing products within 2 months prior to screening
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12-11 (Actual); Primary Completion 2009-03-30 (Actual); Study Completion 2009-03-30 (Actual)

PRIMARY OUTCOMES:
Evidence of safety as determined by assessing adverse events, vital signs, spirometry, ECGs, telemetry, renal biomarkers, safety labs, and physical examination | Part A: 3-4 months; Part B: ~1 month

SECONDARY OUTCOMES:
Plasma or blood concentrations of study drug | Part A: 3-4 months; Part B: ~1 month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 111319 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111319?search=study&search_terms=111319#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111319 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register